CLINICAL TRIAL: NCT01897974
Title: Revisiting Survey Investigating Why Patients Are Not Receiving Home Anti-convulsant Medication Prior to Surgery/or Procedure Involving General Anesthesia
Status: Completed | Type: Observational
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Assistant Clinical Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00276
Record Dates: First submitted 2013-06-26; First posted 2013-07-12 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Seizure disorder: Patients that are on medications for seizure disorder.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Families complete survey to measure medication compliance.

SUMMARY:
Children with seizure disorder face unique challenges during the perioperative period. Fasting, sleep-deprivation, and missed doses of medications while patients are required to have nothing per mouth (NPO) are a few factors that decrease the seizure threshold. The incidence of seizures in this population is unknown but correlated with patient's underlying condition and missed doses of anti-convulsant. Previous work has determined this is not a unique problem.

The investigators initially found compliance extremely poor at 60%. The investigators have made improvement to about 80% compliance through various interventions: education of nursing, availability of anticonvulsant intravenous dosing alternatives, and re-wording the hospital NPO policy. The investigators feel that a new, more focused, survey will help identify, perioperative reasons for non-compliance on part of the parents. This information will be utilized to guide further interventions aimed at improving compliance.

ELIGIBILITY:
Inclusion Criteria:

* We plan to include all children 0-18 years of age on anticonvulsant(s) for seizure disorder.

Exclusion Criteria:

* None.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are taking anti-seizure medications.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Anticonvuslant compliance | 1 Day
  Patients/parents will be asked to complete a questionnaire about whether they took their anticonvulsant the morning of surgery and if not, why not.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States